CLINICAL TRIAL: NCT03164928
Title: A Phase 3 Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Safety and Efficacy of Denosumab in Pediatric Subjects With Glucocorticoid-induced Osteoporosis
Brief Title: Safety and Efficiency of Denosumab in Pediatric Subjects With Glucocorticoid-induced Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20140444; 2016-003083-39 (EudraCT Number)
Record Dates: First submitted 2017-05-08; First posted 2017-05-24 (Actual); Results first posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Evaluate the Safety and Efficacy of Denosumab in Pediatric Subjects With; Glucocorticoid-induced Osteoporosis
Keywords: Denosumab; Pediatric GIOP; Glucocorticoid-induced; Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Other): SC Q6M placebo
  Interventions: Other: Placebo
- Denosumab (Experimental): 1 mg/kg BW (up to a maximum of 60 mg) SC Q6M
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Denosumab — 1mg/kg BW (up to a maximum of 60 mg) SC Q6M
  Arms: Denosumab
Other: Placebo — SC Q6M placebo
  Arms: Placebo

SUMMARY:
To evaluate the effect of denosumab on lumbar spine bone mineral density (BMD) Z-score as assessed by dual-energy X-ray absorptiometry (DXA) at 12 months in children 5 to 17 year of age with Glucocorticoid (GC)-induced osteoporosis (GiOP).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, age 5 to 17 years, inclusive, at the time of informed consent.
* Clinical diagnosis of GiOP as defined by the following (and consistent with the International Society for Clinical Densitometry definition of osteoporosis in children and adolescents [Bishop et al, 2014])
* A confirmed diagnosis of non-malignant condition(s) requiring treatment with systemic GC (including, but not limited to, chronic rheumatologic, gastrointestinal, neurologic, respiratory, and/or nephrological conditions)
* Subjects who are on systemic GC only as replacement therapy for adrenal insufficiency are not eligible for the study - Treatment with systemic GC (intravenous or oral) of any duration for the underlying non-malignant condition(s) within the 12 months prior to screening
* Evidence of at least 1 vertebral compression fracture of Genant grade 1 or higher, as assessed by the central imaging vendor on lateral spine X-rays performed at screening or within 2 months prior to screening; OR, in the absence of vertebral compression fractures, presence of both clinically significant fracture history (ie, ≥ 2 long-bone fractures by age 10 years or ≥ 3 long-bone fractures at any age up to 17 years) and lumbar spine BMD Z-score ≤ -2.0, as assessed by the central imaging vendor.

  • Subject's legally acceptable representative has provided informed consent when the subject is legally too young to provide informed consent and the subject has provided assent based on local regulations and/or guidelines prior to any study-specific activities/procedures being initiated
* A confirmed diagnosis of non-malignant condition(s) requiring treatment with systemic GC (including, but not limited to, chronic rheumatologic, gastrointestinal, neurologic, respiratory, and/or nephrological conditions)
* Subjects who are on systemic GC only as replacement therapy for adrenal insufficiency are not eligible for the study
* Treatment with systemic GC (intravenous or oral) of any duration for the underlying non malignant condition(s) within the 12 months prior to screening
* Prepubertal children should be expected to require significant GC use during the study, per investigator opinion

Exclusion criteria will include the following:

* Current hyperthyroidism (unless well controlled on stable antithyroid therapy)
* Current clinical hypothyroidism (unless well controlled on stable thyroid replacement therapy)
* History of hyperparathyroidism
* Current hypoparathyroidism
* Duchenne muscular dystrophy with symptomatic cardiac abnormality
* Current malabsorption
* Active infection or history of infections
* History of malignancy

  * Any causes of primary or secondary osteoporosis (other than GC use), or previous exposure to non-GC medications, which the investigator considers to have been a major factor contributing to the patient's fracture(s)
  * Current adrenal insufficiency as the sole indication for GC therapy
  * Duchenne muscular dystrophy with symptomatic cardiac abnormality
  * Current malabsorption (in children with serum albumin -lower limit of normal [LLN], malabsorption should be clinically ruled out by the investigator to confirm eligibility)
  * Known intolerance to calcium or vitamin D supplements
  * Active infection or history of infections, defined as follows:
* Any active infection for which systemic anti-infectives were used within 4 weeks prior to screening
* Serious infection, defined as requiring hospitalization or intravenous anti infectives within 8 weeks prior to screening
* Recurrent or chronic infection or other active infection that, in the opinion of the investigator, might compromise the safety of the subject

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2023-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (38):
- United States (6):
  - Childrens Hospital of Los Angeles, Los Angeles, California
  - AI Dupont Hospital for Children, Wilmington, Delaware
  - Indiana University Hospital, Indianapolis, Indiana
  - University of Minnesota Masonic Childrens Hospital Discovery Clinic, Minneapolis, Minnesota
  - Metrohealth Medical Center, Cleveland, Ohio
  - Nationwide Childrens Hospital, Columbus, Ohio
- Perth Childrens Hospital, Nedlands, Western Australia, Australia
- Cliniques Universtaire Saint Luc Universite Catholique de Louvain, Brussels, Belgium
- Medical Centre Synexus Sofia EOOD, Sofia, Bulgaria
- Canada (2):
  - Childrens Hospital of Eastern Ontario, Ottawa, Ontario
  - Centre Hospitalier Universitaire Sainte Justine, Montreal, Quebec
- Colombia (3):
  - Center for Clinical and Basic Research Colombia, Medellín, Antioquia
  - Solano y Terront Servicios Medicos Ltda - Unidad Integral de Endocrinologia Uniendo, Bogota, Cundinamarca
  - Foscal Internacional-Fundacion Oftalmologica de Santander, Floridablanca, Santander Department
- India (4):
  - Gandhi Medical College, Hyderabad, Andhra Pradesh
  - KLES Dr Prabhakar Kore Hospital and Medical Research Centre, Belagavi, Karnataka
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - Christian Medical College, Vellore, Tamil Nadu
- Italy (3):
  - Azienda Ospedaliera Universitaria Meyer, Florence
  - Istituto Auxologico Italiano Istituto di Ricovero e Cura a Carattere Scientifico, Milan
  - Azienda Ospedaliera Policlinico Umberto I, Roma
- RM Pharma Specialists SA de CV, Mexico City, Mexico
- Peru (5):
  - Instituto Nacional de Salud del Nino, Breña, Lima region
  - Centro Especializado de Enfermedades Neoplasicas, Arequipa
  - Hospital Nacional Alberto Sabogal Sologuren, Callao
  - Clinica Angloamericana, Lima
  - Centro de Investigacion Ricardo Palma, Lima
- Russia (4):
  - FSAI Scientific Center of Childrens Health of MoH of the RF, Moscow
  - SBEI of HPE First Moscow state medical university na I M Sechenov of MoH of Russian Federation, Moscow
  - SBHI of Novosibirsk region City Pediatric Clinical Hospital of Emergency Care, Novosibirsk
  - LLC Medical Technologies, Saint Petersburg
- Turkey (Türkiye) (4):
  - Ankara Universitesi Tip Fakultesi, Ankara
  - Ataturk Universitesi Tip Fakultesi, Erzurum
  - Marmara Universitesi Pendik Egitim Arastirma Hastanesi, Istanbul
  - Ege Universitesi Tip Fakultesi, Izmir
- Ukraine (3):
  - CI Dnipropetrovsk Regional Children Clinical Hospital of Dnipropetrovsk Regional Council, Dnipro
  - Communal Institution of Healthcare Kharkiv City Clinical Children Hospital 16, Kharkiv
  - National Childrens Specialized Hospital OHMATDYT, Kyiv

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 12 center(s) in Australia, Canada, Columbia, India, Peru, Russia, Turkey, Ukraine, and the United States between May 2018 and December 2023.
Pre-assignment Details: Participants were randomized in a 2:1 allocation ratio to receive either denosumab or placebo respectively, in a double-blind manner during the 12-month placebo-controlled double-blind Treatment Period. This was followed by a 12-month denosumab Open-label Treatment Period and a 12-month Off-treatment Observation Period.
Groups:
- Denosumab/Denosumab: Participants received 1 mg/kg Denosumab by SC injection up to a maximum of 60 mg, Q6M for 24 months during the Treatment Period. Participants were then followed for an additional 12 months during the Off-treatment Observation Period.
- Placebo/Denosumab: Participants received matching placebo by SC injection Q6M for the first 12 months of the Treatment Period. This was followed by 1 mg/kg Denosumab administered by SC injection, up to a maximum of 60 mg, Q6M for the second 12 months of the Treatment Period. Participants were then followed for an additional 12 months during the Off-treatment Observation Period.
Period: Overall Study
Arm/Group | Denosumab/Denosumab | Placebo/Denosumab
Started | 16 | 8
Completed | 15 | 8
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): all participants enrolled into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Denosumab/Denosumab | Placebo/Denosumab | Total
Number analyzed (Participants) | 16 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 13.8 (2.3) | 12.8 (2.1) | 13.4 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 10 | 4 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 15 | 5 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 5 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Bone Mineral Density (BMD) Z-score at Baseline [Mean (Standard Deviation); unit: Z-score] — BMD was assessed by DXA and results were converted to z-scores, indicating number of standard deviations from the reference population's mean, with 0 denoting the mean. Population: Only participants with available data have been included.
  Z-score
    Lumbar Spine | -1.95 (1.03) | -3.60 (1.77) | -2.50 (1.51)
    Total Hip: number analyzed (Participants) | 16 | 7 | 23
    Total Hip | -3.14 (1.70) | -4.56 (2.08) | -3.58 (1.90)
    Femoral Neck: number analyzed (Participants) | 16 | 7 | 23
    Femoral Neck | -3.35 (1.91) | -4.78 (2.80) | -3.79 (2.25)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Lumbar Spine BMD Z-score as Assessed by Dual-energy X-ray Absorptiometry (DXA) at 12 Months
Description: Lumbar spine BMD was assessed by DXA and analyzed by analysis of covariance (ANCOVA) including treatment (denosumab vs placebo), baseline age, and baseline BMD z-score. DXA results were converted to z-scores, indicating number of standard deviations from the reference population's mean, with 0 denoting the mean. Positive changes from baseline signify lumbar spine BMD improvement.
Time Frame: Baseline and 12 Months
Population: Primary DXA Analysis Set: all participants in the FAS with baseline and ≥ 1 postbaseline valid DXA assessment of lumbar spine provided by the central imaging vendor during the first 12 months.
Measure: Least Squares Mean (95% Confidence Interval); unit: Z-score
Arm/Group | Denosumab/Denosumab | Placebo/Denosumab
Number analyzed (Participants) | 15 | 8
Z-score | 0.23 [-0.054 to 0.506] | 0.11 [-0.304 to 0.532]
Statistical Analysis 1: Comparison: Denosumab/Denosumab vs Placebo/Denosumab; Test type: Superiority; p = 0.68, ANCOVA; Least Squares Mean Difference = 0.11, 95% CI 2-sided [-0.450 to 0.673]

2. Secondary Outcome: Change From Baseline in Lumbar Spine BMD Z-score as Assessed by DXA at 6, 18, 24, and 36 Months
Description: Lumbar spine BMD was assessed by DXA and analyzed by repeated measures analysis with randomization group, visit, baseline age, and baseline BMD z-score as fixed effects. Treatment-by-visit was included as an interaction term. DXA results were converted to z-scores, indicating number of standard deviations from the reference population's mean, with 0 denoting the mean. Positive changes from baseline signify lumbar spine BMD improvement.
Time Frame: Baseline and 6, 18, 24, and 36 Months
Population: DXA Analysis Set: all participants in the FAS with baseline and ≥ 1 postbaseline valid DXA assessment for lumbar spine as provided by the central imaging vendor. All participants included in the Overall Number of Participants Analyzed contributed data to this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: Z-score
Arm/Group | Denosumab/Denosumab | Placebo/Denosumab
Number analyzed (Participants) | 15 | 8
Z-score
  Month 6: number analyzed (Participants) | 14 | 6
  Month 6 | 0.28 [0.095 to 0.468] | 0.11 [-0.176 to 0.391]
  Month 18: number analyzed (Participants) | 15 | 7
  Month 18 | 0.32 [-0.034 to 0.679] | 0.30 [-0.206 to 0.800]
  Month 24: number analyzed (Participants) | 13 | 7
  Month 24 | 0.37 [-0.017 to 0.755] | 0.26 [-0.285 to 0.801]
  Month 36: number analyzed (Participants) | 9 | 5
  Month 36 | -0.23 [-0.833 to 0.372] | 0.57 [-0.268 to 1.416]
Statistical Analysis 1: Comparison: Denosumab/Denosumab vs Placebo/Denosumab; Month 6; Test type: Superiority; p = 0.34, Repeated Measures Model; Least Squares Mean Difference = 0.17, 95% CI 2-sided [-0.194 to 0.542]
Statistical Analysis 2: Comparison: Denosumab/Denosumab vs Placebo/Denosumab; Month 18; Test type: Superiority; p = 0.93, Repeated Measures Model; Least Squares Mean Difference = 0.03, 95% CI 2-sided [-0.609 to 0.661]
Statistical Analysis 3: Comparison: Denosumab/Denosumab vs Placebo/Denosumab; Month 24; Test type: Superiority; p = 0.74, Repeated Measures Model; Least Squares Mean Difference = 0.11, 95% CI 2-sided [-0.572 to 0.795]
Statistical Analysis 4: Comparison: Denosumab/Denosumab vs Placebo/Denosumab; Month 36; Test type: Superiority; p = 0.12, Repeated Measures Model; Least Squares Means Difference = -0.80, 95% CI 2-sided [-1.848 to 0.239]

3. Secondary Outcome: Change From Baseline in Proximal Femur BMD Z-score as Assessed by DXA at 6, 12, 18, 24, and 36 Months
Description: Proximal femur (total hip and femoral neck) BMD was assessed by DXA and analyzed by repeated measures analysis with randomization group, visit, baseline age, and baseline BMD z-score as fixed effects. Treatment-by-visit was included as an interaction term. DXA results were converted to z-scores, indicating number of standard deviations from the reference population's mean, with 0 denoting the mean. Positive changes from baseline signify proximal femur BMD improvement.
Time Frame: Baseline and 6, 12, 18, 24, and 36 Months
Population: DXA Analysis Set: all participants in the FAS with baseline and ≥ 1 postbaseline valid DXA assessment for total hip and femoral neck as provided by the central imaging vendor.
Measure: Least Squares Mean (95% Confidence Interval); unit: Z-score
Arm/Group | Denosumab/Denosumab | Placebo/Denosumab
Number analyzed (Participants) | 15 | 7
Z-score
  Month 6 (Total Hip): number analyzed (Participants) | 13 | 5
  Month 6 (Total Hip) | 0.22 [-0.103 to 0.552] | 0.64 [0.104 to 1.171]
  Month 12 (Total Hip): number analyzed (Participants) | 14 | 7
  Month 12 (Total Hip) | 0.24 [-0.079 to 0.554] | 0.30 [-0.168 to 0.759]
  Month 18 (Total Hip): number analyzed (Participants) | 15 | 6
  Month 18 (Total Hip) | 0.48 [0.015 to 0.937] | 0.75 [0.061 to 1.434]
  Month 24 (Total Hip): number analyzed (Participants) | 13 | 6
  Month 24 (Total Hip) | 0.52 [0.000 to 1.033] | 0.69 [-0.062 to 1.447]
  Month 36 (Total Hip): number analyzed (Participants) | 9 | 5
  Month 36 (Total Hip) | 0.64 [-0.149 to 1.436] | 0.73 [-0.384 to 1.850]
  Month 6 (Femoral Neck): number analyzed (Participants) | 13 | 5
  Month 6 (Femoral Neck) | 0.42 [0.000 to 0.849] | 0.60 [-0.037 to 1.241]
  Month 12 (Femoral Neck): number analyzed (Participants) | 14 | 7
  Month 12 (Femoral Neck) | 0.53 [0.029 to 1.030] | 0.43 [-0.294 to 1.161]
  Month 18 (Femoral Neck): number analyzed (Participants) | 15 | 6
  Month 18 (Femoral Neck) | 0.85 [0.261 to 1.446] | 0.48 [-0.387 to 1.350]
  Month 24 (Femoral Neck): number analyzed (Participants) | 13 | 6
  Month 24 (Femoral Neck) | 0.75 [0.000 to 1.495] | 0.64 [-0.449 to 1.724]
  Month 36 (Femoral Neck): number analyzed (Participants) | 9 | 5
  Month 36 (Femoral Neck) | 1.00 [-0.008 to 2.012] | 0.63 [-0.798 to 2.050]
Statistical Analysis 1: Comparison: Denosumab/Denosumab vs Placebo/Denosumab; Month 6 (Total Hip); Test type: Superiority; p = 0.19, Repeated Measures Model; Least Squares Mean Difference = -0.41, 95% CI 2-sided [-1.050 to 0.223]
Statistical Analysis 2: Comparison: Denosumab/Denosumab vs Placebo/Denosumab; Month 12 (Total Hip); Test type: Superiority; p = 0.83, Repeated Measures Model; Least Squares Mean Difference = -0.06, 95% CI 2-sided [-0.631 to 0.515]
Statistical Analysis 3: Comparison: Denosumab/Denosumab vs Placebo/Denosumab; Month 18 (Total Hip); Test type: Superiority; p = 0.51, Repeated Measures Model; Least Squares Mean Difference = -0.27, 95% CI 2-sided [-1.108 to 0.565]
Statistical Analysis 4: Comparison: Denosumab/Denosumab vs Placebo/Denosumab; Month 24 (Total Hip); Test type: Superiority; p = 0.69, Repeated Measures Model; Least Squares Mean Difference = -0.18, 95% CI 2-sided [-1.098 to 0.746]
Statistical Analysis 5: Comparison: Denosumab/Denosumab vs Placebo/Denosumab; Month 36 (Total Hip); Test type: Superiority; p = 0.89, Repeated Measures Model; Least Squares Mean Difference = -0.09, 95% CI 2-sided [-1.465 to 1.286]
Statistical Analysis 6: Comparison: Denosumab/Denosumab vs Placebo/Denosumab; Month 6 (Femoral Neck); Test type: Superiority; p = 0.64, Repeated Measures Model; Least Squares Mean Difference = -0.18, 95% CI 2-sided [-0.969 to 0.614]
Statistical Analysis 7: Comparison: Denosumab/Denosumab vs Placebo/Denosumab; Month 12 (Femoral Neck); Test type: Superiority; p = 0.83, Repeated Measures Model; Least Squares Mean Difference = 0.10, 95% CI 2-sided [-0.808 to 1.000]
Statistical Analysis 8: Comparison: Denosumab/Denosumab vs Placebo/Denosumab; Month 18 (Femoral Neck); Test type: Superiority; p = 0.48, Repeated Measures Model; Least Squares Mean Difference = 0.37, 95% CI 2-sided [-0.697 to 1.442]
Statistical Analysis 9: Comparison: Denosumab/Denosumab vs Placebo/Denosumab; Month 24 (Femoral Neck); Test type: Superiority; p = 0.86, Repeated Measures Model; Least Squares Mean Difference = 0.11, 95% CI 2-sided [-1.222 to 1.443]
Statistical Analysis 10: Comparison: Denosumab/Denosumab vs Placebo/Denosumab; Month 36 (Femoral Neck); Test type: Superiority; p = 0.66, Repeated Measures Model; Least Squares Mean Difference = 0.38, 95% CI 2-sided [-1.378 to 2.130]

4. Secondary Outcome: Number of Participants With X-ray Confirmed Long-bone Fractures and/or Vertebral Fractures at 12, 24, and 36 Months
Description: Number of participants who have at least one long bone fracture or vertebral fracture, and number of participants who have more than one long bone fracture or vertebral fracture.
Time Frame: Month 12, 24, and 36
Population: FAS: all participants randomized into the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Denosumab/Denosumab | Placebo/Denosumab
Number analyzed (Participants) | 16 | 8
Participants
  Month 12 (at least 1 fracture) | 2 | 2
  Month 24 (at least 1 fracture) | 3 | 3
  Month 36 (at least 1 fracture) | 3 | 3
  Month 12 (more than 1 fracture) | 2 | 1
  Month 24 (more than 1 fracture) | 2 | 0
  Month 36 (more than 1 fracture) | 3 | 1

5. Secondary Outcome: Number of Participants With Improving Vertebral Fractures at 12, 24, and 36 Months
Description: Number of participants with improving vertebral fractures. An improving fracture is defined as one showing signs of healing/repair from baseline as assessed by X-ray.
Time Frame: Month 12, 24, and 36
Population: Vertebral Fracture Analysis Set: all participants in the FAS who have a non-missing baseline and ≥ 1 non-missing postbaseline X-ray vertebral evaluation as provided by the central imaging vendor, on or before the time point under consideration.
Measure: Count of Participants; unit: Participants
Arm/Group | Denosumab/Denosumab | Placebo/Denosumab
Number analyzed (Participants) | 15 | 7
Participants
  Month 12 | 3 | 1
  Month 24 | 2 | 1
  Month 36 | 1 | 2

6. Secondary Outcome: Number of Participants With New and Worsening Vertebral and Non-vertebral Fractures at 12, 24, and 36 Months
Description: Number of participants who have at least one vertebral fracture or non-vertebral fracture, and number of participants who have more than one vertebral fracture or non-vertebral fracture.
Time Frame: Month 12, 24, and 36
Population: FAS: all participants randomized into the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Denosumab/Denosumab | Placebo/Denosumab
Number analyzed (Participants) | 16 | 8
Participants
  Month 12 (at least 1 fracture) | 2 | 2
  Month 24 (at least 1 fracture) | 3 | 3
  Month 36 (at least 1 fracture) | 3 | 3
  Month 12 (more than 1 fracture) | 2 | 1
  Month 24 (more than 1 fracture) | 2 | 0
  Month 36 (more than 1 fracture) | 3 | 1

7. Secondary Outcome: Change From Baseline in Child Health Questionnaire-Parent Form-50 (CHQ-PF-50) Physical Summary Score at 12, 24, and 36 Months
Description: The CHQ-PF-50 is a 50-item questionnaire to be completed by the parents or guardians of children between 5 and 18 years of age. The physical summary score ranges from 0-100 with higher scores indicating better physical health.
Time Frame: Baseline and month 12, 24, and 36
Population: Patient Reported Outcomes (PRO) Analysis Set: all participants in the FAS with baseline and at least one valid CHQ-PF-50 response at post-baseline. All participants included in the Overall Number of Participants Analyzed contributed data to this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Denosumab/Denosumab | Placebo/Denosumab
Number analyzed (Participants) | 14 | 7
Scores on a scale
  Month 12: number analyzed (Participants) | 12 | 7
  Month 12 | 5.26 (8.88) | 8.53 (16.39)
  Month 24: number analyzed (Participants) | 13 | 5
  Month 24 | 5.62 (7.39) | 19.88 (15.20)
  Month 36: number analyzed (Participants) | 9 | 5
  Month 36 | 4.48 (8.89) | 14.18 (8.14)

8. Secondary Outcome: Change From Baseline in CHQ-PF-50 Psychological Summary Score at 12, 24, and 36 Months
Description: The CHQ-PF-50 is a 50-item questionnaire to be completed by the parents or guardians of children between 5 and 18 years of age. The psychological summary score ranges from 0-100 with higher scores indicating better psychological health.
Time Frame: Baseline and Month 12, 24, and 36
Population: PRO Analysis Set: all participants in the FAS with baseline and at least one valid CHQ-PF-50 response at post-baseline. All participants included in the Overall Number of Participants Analyzed contributed data to this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Denosumab/Denosumab | Placebo/Denosumab
Number analyzed (Participants) | 14 | 7
Scores on a scale
  Month 12: number analyzed (Participants) | 12 | 7
  Month 12 | 0.71 (9.15) | -0.10 (12.52)
  Month 24: number analyzed (Participants) | 13 | 5
  Month 24 | 2.58 (12.58) | 1.90 (9.76)
  Month 36: number analyzed (Participants) | 9 | 5
  Month 36 | 5.20 (10.09) | 2.00 (9.33)

9. Secondary Outcome: Change From Baseline in Childhood Health Assessment Questionnaire (CHAQ) Disability Index Score at 12, 24, and 36 Months
Description: The CHAQ was developed to measure the physical functioning in children 6 months to 18 years of age. It consists of 54 questions related to the child's ability to perform various activities of daily living. Depending on the question asked, each question is scored either 0 to 3 based on the level of difficulty experienced by the child or 0-1 based on whether the child required assistance from another person or used an aid or other device. All CHAQ questions were scored and converted to a total index score ranging from 0-3, where higher scores indicate greater disability.
Time Frame: Baseline and Month 12, 24, and 36
Population: PRO Analysis Set: all participants in the FAS with baseline and at least one valid CHAQ response at post-baseline. All participants included in the Overall Number of Participants Analyzed contributed data to this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Denosumab/Denosumab | Placebo/Denosumab
Number analyzed (Participants) | 14 | 7
Scores on a scale
  Month 12: number analyzed (Participants) | 12 | 7
  Month 12 | -0.06 (0.32) | -0.29 (0.44)
  Month 24: number analyzed (Participants) | 13 | 5
  Month 24 | -0.09 (0.33) | -0.30 (0.49)
  Month 36: number analyzed (Participants) | 8 | 5
  Month 36 | -0.12 (0.45) | -0.43 (0.45)

10. Secondary Outcome: Change From Baseline in Wong-Baker FACES Pain Rating Scale (WBFPRS) at 12, 24, and 36 Months
Description: The WBFPRS is a horizontal pain scale for children 3-18 years which consists of 6 faces that range from a smiling "no hurt" face with a score of 0 to a crying "hurts worst" face with a score of 10.
Time Frame: Baseline and Month 12, 24, and 36
Population: PRO Analysis Set: all participants in the FAS with baseline and at least one valid WBFPRS response at post-baseline. All participants included in the Overall Number of Participants Analyzed contributed data to this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Denosumab/Denosumab | Placebo/Denosumab
Number analyzed (Participants) | 14 | 7
Scores on a scale
  Month 12: number analyzed (Participants) | 11 | 7
  Month 12 | -0.7 (3.3) | -0.3 (3.9)
  Month 24: number analyzed (Participants) | 13 | 5
  Month 24 | -0.6 (2.9) | -2.4 (0.9)
  Month 36: number analyzed (Participants) | 8 | 5
  Month 36 | -2.5 (1.8) | 0.0 (1.4)

11. Secondary Outcome: Change From Baseline in Growth Velocity Z-score (Height) at 12, 24, and 36 Months
Description: Growth velocity was determined by calculating age-adjusted z-scores for height, weight, and body mass index (BMI). Z-scores represent the number of standard deviations from the reference population's mean, with 0 denoting the mean. Positive changes from baseline signify increased growth velocity.
Time Frame: Baseline and Month 12, 24, and 36
Population: Growth Velocity Analysis Set: all participants in the FAS who have non-missing height and age in total months at baseline and postbaseline. Only participants with available data for growth velocity (height) are included. All participants included in the Overall Number of Participants Analyzed contributed data to this outcome measure.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Denosumab/Denosumab | Placebo/Denosumab
Number analyzed (Participants) | 15 | 8
Z-score
  Month 12: number analyzed (Participants) | 13 | 8
  Month 12 | -0.18 (0.46) | -0.07 (0.84)
  Month 24: number analyzed (Participants) | 12 | 7
  Month 24 | -0.11 (0.90) | -0.27 (1.17)
  Month 36: number analyzed (Participants) | 12 | 7
  Month 36 | -0.33 (0.84) | 0.01 (1.35)

12. Secondary Outcome: Change From Baseline in Growth Velocity Z-score (Weight) at 12, 24, and 36 Months
Description: Growth velocity was determined by calculating age-adjusted z-scores for height, weight, and BMI. Z-scores represent the number of standard deviations from the reference population's mean, with 0 denoting the mean. Positive changes from baseline signify increased growth velocity.
Time Frame: Baseline and Month 12, 24, and 36
Population: Growth Velocity Analysis Set: all participants in the FAS who have non-missing weight and age in total months at baseline and postbaseline. Only participants with available data for growth velocity (weight) are included.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Denosumab/Denosumab | Placebo/Denosumab
Number analyzed (Participants) | 16 | 8
Z-score
  Month 12: number analyzed (Participants) | 15 | 8
  Month 12 | -0.12 (0.44) | -0.10 (0.49)
  Month 24: number analyzed (Participants) | 12 | 7
  Month 24 | -0.22 (0.73) | -0.68 (0.62)
  Month 36: number analyzed (Participants) | 12 | 7
  Month 36 | -0.32 (0.90) | -0.44 (0.60)

13. Secondary Outcome: Change From Baseline in Growth Velocity Z-score (BMI) at 12, 24, and 36 Months
Description: as for outcome 12
Time Frame: Baseline and Month 12, 24, and 36
Population: Growth Velocity Analysis Set: all participants in the FAS who have non-missing BMI and age in total months at baseline and postbaseline. Only participants with available data for growth velocity (BMI) are included. All participants included in the Overall Number of Participants Analyzed contributed data to this outcome measure.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Denosumab/Denosumab | Placebo/Denosumab
Number analyzed (Participants) | 15 | 8
Z-score
  Month 12: number analyzed (Participants) | 13 | 8
  Month 12 | -0.03 (0.53) | -0.14 (0.54)
  Month 24: number analyzed (Participants) | 12 | 7
  Month 24 | -0.12 (0.80) | -0.75 (1.02)
  Month 36: number analyzed (Participants) | 12 | 7
  Month 36 | -0.12 (0.84) | -0.72 (0.97)

14. Secondary Outcome: Mean Serum Concentration of Denosumab
Time Frame: Day 1, Day 10, Day 30, Month 3, Month 6, Month 12, and Month 18
Population: PK Analysis Set: all participants in the FAS who have ≥ 1 denosumab reported result.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Denosumab/Denosumab | Placebo/Denosumab
Number analyzed (Participants) | 15 | 8
ng/mL
  Day 1: number analyzed (Participants) | 14 | 0
  Day 1 | 0.00 (0.00) |
  Day 10: number analyzed (Participants) | 11 | 0
  Day 10 | 10300 (7900) |
  Day 30: number analyzed (Participants) | 9 | 0
  Day 30 | 6830 (4770) |
  Month 3: number analyzed (Participants) | 10 | 0
  Month 3 | 1100 (935) |
  Month 6: number analyzed (Participants) | 12 | 0
  Month 6 | 141 (338) |
  Month 12: number analyzed (Participants) | 11 | 7
  Month 12 | 157 (349) | 0.00 (0.00)
  Month 18: number analyzed (Participants) | 12 | 8
  Month 18 | 49 (154) | 7.61 (21.5)

ADVERSE EVENTS:
Time Frame: From date of enrollment through last dose, up to 36 months.
Groups:
- Baseline-Month 12: Placebo: Participants received placebo by SC injection during the first 12 months of the Treatment Period.
- Baseline-Month 12: Denosumab: Participants received 1 mg/kg Denosumab up to a maximum of 60 mg, Q6M by SC injection during the first 12 months of the Treatment Period.
- Baseline-Month 24: Placebo/Denosumab: Participants received matching placebo by SC injection Q6M for the first 12 months of the Treatment Period. This was followed by 1 mg/kg Denosumab administered by SC injection Q6M for the second 12 months of the Treatment Period.
- Baseline-Month 24: Denosumab/Denosumab: Participants received 1 mg/kg Denosumab by SC injection up to a maximum of 60 mg, Q6M for 24 months during the Treatment Period.
- Baseline-Month 36: Placebo/Denosumab: Participants received matching placebo by SC injection Q6M for the first 12 months of the Treatment Period. This was followed by 1 mg/kg Denosumab up to a maximum of 60 mg, Q6M administered by SC injection for the second 12 months of the Treatment Period. Participants were then followed for an additional 12 months during the Off-treatment Observation Period.
- Baseline-Month 36: Denosumab/Denosumab: Participants received 1 mg/kg Denosumab by SC injection up to a maximum of 60 mg, Q6M for 24 months during the Treatment Period. Participants were then followed for an additional 12 months during the Off-treatment Observation Period.
Arm/Group | Baseline-Month 12: Placebo | Baseline-Month 12: Denosumab | Baseline-Month 24: Placebo/Denosumab | Baseline-Month 24: Denosumab/Denosumab | Baseline-Month 36: Placebo/Denosumab | Baseline-Month 36: Denosumab/Denosumab
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/16 | 0/8 | 0/16 | 0/8 | 0/16
Serious Adverse Events (participants affected / at risk) | 1/8 | 3/16 | 1/8 | 3/16 | 2/8 | 4/16
Other Adverse Events (participants affected / at risk) | 5/8 | 11/16 | 5/8 | 12/16 | 5/8 | 13/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Baseline-Month 12: Placebo (N=8) | Baseline-Month 12: Denosumab (N=16) | Baseline-Month 24: Placebo/Denosumab (N=8) | Baseline-Month 24: Denosumab/Denosumab (N=16) | Baseline-Month 36: Placebo/Denosumab (N=8) | Baseline-Month 36: Denosumab/Denosumab (N=16)
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 1 | 0 | 1 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Brain contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Baseline-Month 12: Placebo (N=8) | Baseline-Month 12: Denosumab (N=16) | Baseline-Month 24: Placebo/Denosumab (N=8) | Baseline-Month 24: Denosumab/Denosumab (N=16) | Baseline-Month 36: Placebo/Denosumab (N=8) | Baseline-Month 36: Denosumab/Denosumab (N=16)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 2 | 0 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 2 | 0 | 2
Intracranial lipoma (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0
Delayed puberty (Endocrine disorders) | 0 | 1 | 0 | 1 | 0 | 2
Astigmatism (Eye disorders) | 1 | 0 | 1 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 1
Cataract subcapsular (Eye disorders) | 1 | 0 | 1 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 0
Duodenal bulb deformity (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Duodenogastric reflux (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0 | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 0 | 1 | 0 | 1
Hyperthermia (General disorders) | 1 | 0 | 1 | 0 | 1 | 0
Injection site pain (General disorders) | 0 | 1 | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 1 | 0 | 2
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Biliary tract disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Balanitis candida (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 1
COVID-19 pneumonia (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0
Chronic tonsillitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1
Coronavirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Epstein-Barr virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1
Gingivitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 3
Respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1
Skin infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1
Varicella (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1
Viral tonsillitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1
Vulvitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Bone density decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Autoimmune arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2 | 0 | 2
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dwarfism (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 2 | 1 | 2 | 1 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myelopathy (Nervous system disorders) | 1 | 0 | 1 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 1
Metabolic nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Central sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1 | 0
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chronic spontaneous urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/28/NCT03164928/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-12): https://cdn.clinicaltrials.gov/large-docs/28/NCT03164928/SAP_001.pdf